CLINICAL TRIAL: NCT03227861
Title: A Phase 3, Single-arm, Open-label Study to Evaluate the Efficacy and Safety of Darunavir/ Cobicistat/ Emtricitabine/ Tenofovir Alafenamide (D/C/F/TAF) Once Daily Fixed-dose Combination (FDC) Regimen in Newly Diagnosed, Antiretroviral Treatment-naïve Human Immunodeficiency Virus Type 1 (HIV-1) Infected Subjects Receiving Care in a Test and Treat Model of Care
Brief Title: A Study to Evaluate the Efficacy and Safety of (D/C/F/TAF) Once Daily Fixed Dose Combination (FDC) Regimen in Newly Diagnosed, Antiretroviral Treatment-naive Human Immunodeficiency Virus Type 1 (HIV-1) Infected Participants Receiving Care in a Test and Treat Model of Care
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR108345; TMC114FD2HTX3002 (Other: Janssen Scientific Affairs, LLC)
Record Dates: First submitted 2017-07-21; First posted 2017-07-24 (Actual); Results first posted 2020-01-07 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: HIV-1
MeSH Terms: interventions — Racivir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- DRV 800 mg + COBI 150 mg + FTC 200 mg + TAF 10 mg FDC (Experimental): Participants will receive oral tablet containing Darunavir 800 milligram (mg)/ Cobicistat 150 mg/ Emtricitabine 200 mg/ Tenofovir Alafenamide 10 mg (D/C/F/TAF) fixed-dose combination (FDC) once daily within 24 hours of the screening/baseline visit.
  Interventions: Drug: DRV 800 mg + COBI 150 mg + FTC 200 mg + TAF 10 mg FDC

INTERVENTIONS:
Drug: DRV 800 mg + COBI 150 mg + FTC 200 mg + TAF 10 mg FDC — Participants will receive oral tablet containing D 800 mg /C 150 mg /F 200 mg /TAF 10 mg FDC once daily within 24 hours of the screening/ baseline visit.

SUMMARY:
The purpose of this study is to assess the efficacy of Darunavir/ Cobicistat/ Emtricitabine/ Tenofovir Alafenamide (D/C/F/TAF) fixed-dose combination (FDC) in a Test and Treat model of care in newly diagnosed human immunodeficiency virus (HIV-1)-infected, treatment-naive participants as determined by the proportion of virologic responders defined as having (HIV)-1 ribonucleic acid (RNA) lesser than 50 copies per milliliter (copies/mL) at Week 48.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed with human immunodeficiency virus type 1 (HIV-1) evidenced by any of the following within 2 weeks of the screening/baseline visit: a) HIV Rapid Antibody positive; or b) HIV Immunoassay positive; or c) Positive p24 antigen and a HIV-1 ribonucleic acid (RNA) viral load greater than or equal to (>=) 5,000 copies per milliliter (copies/ mL); or d) Non-reactive HIV-1 antibody/antigen assays and HIV-1 RNA viral load (>=) 5,000 copies/mL. HIV-1 RNA viral load must be confirmed once within 1 week of initial HIV-1 RNA viral load test
* Antiretroviral treatment-naïve, except for the use of TRUVADA® for pre-exposure prophylaxis (PrEP)
* Must be able to swallow whole tablets
* A woman must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during the study and for 90 days after receiving the last dose of study drug
* A woman of childbearing potential must have a negative urine pregnancy test at screening

Exclusion Criteria:

* Known active cryptococcal infection, active toxoplasmic encephalitis, Mycobacterium tuberculosis infection, or another acquired immunodeficiency syndrome (AIDS) -defining condition that in the judgement of the investigator would increase the risk of morbidity or mortality
* Known history of clinically relevant hepatic disease or hepatitis that in the investigator's judgement is not compatible with Darunavir/ Cobicistat/ Emtricitabine/ Tenofovir Alafenamide (D/C/F/TAF FDC)
* Known history of cirrhosis as diagnosed based on local practices
* Known history of chronic ([>=] 3 months) renal insufficiency, defined as having an estimated glomerular filtration rate (eGFR) less than (<) 50 milliliter per minute (mL/min) according to the Modification of Diet in Renal Disease (MDRD) formula
* Pregnant, or breast-feeding, or planning to become pregnant while enrolled in this study or within 90 days after the last dose of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2017-07-31 (Actual); Primary Completion 2019-01-03 (Actual); Study Completion 2019-09-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Scientific Affairs, LLC Clinical Trial, Study Director — Janssen Scientific Affairs, LLC
Locations (16):
- United States (16):
  - Spectrum Medical Group, Phoenix, Arizona
  - The Office of Franco Felizarta, MD, Bakersfield, California
  - Jeffrey Goodman Clinic - DBA Los Angeles Gay and Lesbian Center, Los Angeles, California
  - Whitman Walker Health, Washington D.C., District of Columbia
  - Midway Immunology and Research Center, Ft. Pierce, Florida
  - University of Miami, Miami, Florida
  - Orlando Immunology Center, Orlando, Florida
  - Chatham County Health Department, Savannah, Georgia
  - The Ruth M. Rothstein CORE Center, Chicago, Illinois
  - Saint Michaels Medical Center - Infectious Disease, Newark, New Jersey
  - Southwest CARE Center, Albuquerque, New Mexico
  - Southwest CARE Center, Santa Fe, New Mexico
  - North Texas Infectious Diseases Consultants, Dallas, Texas
  - Texas Centers for Infectious Disease Associates, Fort Worth, Texas
  - Therapeutic Concepts - Donald R Watkins Foundation, Houston, Texas
  - Gordon Crofoot, MD, Houston, Texas

REFERENCES:
- [Derived] Dunn K, Rogers R, Simonson RB, Luo D, Sheng S, Kassam PT, Seyedkazemi S, Hardy H. Rapid initiation of darunavir/cobicistat/emtricitabine/tenofovir alafenamide in acute and early HIV-1 infection: a DIAMOND subgroup analysis. HIV Res Clin Pract. 2021 Apr;22(2):55-61. doi: 10.1080/25787489.2021.1915652. Epub 2021 May 17. PMID 33999786
- [Derived] Huhn GD, Crofoot G, Ramgopal M, Gathe J, Bolan R, Luo D, Simonson RB, Nettles RE, Benson C, Dunn K. Darunavir/Cobicistat/Emtricitabine/Tenofovir Alafenamide in a Rapid-Initiation Model of Care for Human Immunodeficiency Virus Type 1 Infection: Primary Analysis of the DIAMOND Study. Clin Infect Dis. 2020 Dec 15;71(12):3110-3117. doi: 10.1093/cid/ciz1213. PMID 31879782

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Out of 97 participants who completed the main study, 80 participants continued into the extension phase and were treated with Darunavir/Cobicistat/Emtricitabine/Tenofovir alafenamide (D/C/F/TAF) fixed dose combination (FDC).
Groups:
- D/C/F/TAF: Participants received oral tablet containing Darunavir 800 milligram (mg)/Cobicistat 150 mg/Emtricitabine 200 mg/Tenofovir alafenamide 10 mg (D/C/F/TAF) as Fixed-dose Combination (FDC) from Day 1 to Week 48. Participants who completed the Week 48 visit were given the opportunity to continue D/C/F/TAF treatment during the extension phase until the D/C/F/TAF FDC tablet became commercially available and was reimbursed, or could be accessed through another source, or until the sponsor terminated clinical development (Up to 96 Weeks).
Period: Main Study Period (Week 0 to Week 48)
Arm/Group | D/C/F/TAF
Started | 109
Completed | 97
Not Completed | 12
Not completed — Lost to Follow-up | 4
Not completed — Withdrawal by Subject | 1
Not completed — Adverse Event | 1
Not completed — Protocol Violation | 1
Not completed — Other | 5
Period: Extension Period (Week 48 to Week 96)
Arm/Group | D/C/F/TAF
Started | 80 (17 participants were not willing to enter extension study and discontinued after main study.)
Completed | 0
Not Completed | 80
Not completed — Transition to Commercial D/C/F/TAF | 55
Not completed — Transition to Other ARV Treatment | 16
Not completed — Lost to Follow-up | 6
Not completed — Adverse Event | 1
Not completed — Other | 2

BASELINE CHARACTERISTICS:
Groups:
- D/C/F/TAF: Participants received oral tablet containing Darunavir 800 milligram (mg)/Cobicistat 150 mg/Emtricitabine 200 mg/Tenofovir alafenamide 10 mg (D/C/F/TAF) as Fixed-dose Combination (FDC) from Day 1 to Week 48.
Arm/Group | D/C/F/TAF
Number analyzed (Participants) | 109
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.5 (12.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 95
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 35
  White | 65
  More than one race | 3
  Unknown or Not Reported | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 109

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Human Immunodeficiency Virus (HIV)-1 Ribonucleic Acid (RNA) Less Than (<) 50 Copies Per Milliliter (Copies/mL) (Virologic Response) at Week 48 Defined by Food and Drug Administration (FDA) Snapshot Approach
Description: Percentage of participants with a HIV-1 RNA < 50 copies per mL were assessed using FDA snapshot approach which defines a participant's virologic response status using only the viral load at the predefined time point within a window of time, along with study drug discontinuation status. If HIV RNA level is < 50 copies per mL at Week 48, it is considered as virologic success as per the snapshot approach.
Time Frame: Week 48
Population: The intent-to-treat (ITT) analysis set included all the participants who were randomized and received at least one dose of study treatment in the study.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- D/C/F/TAF: Main Study: Participants received oral tablet containing Darunavir 800 milligram (mg)/Cobicistat 150 mg/Emtricitabine 200 mg/Tenofovir alafenamide 10 mg (D/C/F/TAF) as Fixed-dose Combination (FDC) from Day 1 to Week 48.
Arm/Group | D/C/F/TAF: Main Study
Number analyzed (Participants) | 109
Percentage of participants | 84.4 [76.44 to 90.03]

2. Secondary Outcome: Change From Baseline in log10 HIV-1 RNA Viral Load (<50/200 Copies/mL) at Weeks 2, 4, 8, 12, 24, 36, and 48
Description: Change from baseline in log10 HIV-1 RNA viral load (<50/200 copies/mL) at Weeks 2, 4, 8, 12, 24, 36, and 48 were reported.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 24, 36, and 48
Population: The ITT analysis set included all participants who were randomized and received at least one dose of study treatment in study. Here, n (number analyzed) signifies participants analyzed for this outcome measure (OM) at specified timepoints.
Measure: Mean (Standard Error); unit: log10 HIV-1 RNA copies per mL
Arm/Group | D/C/F/TAF: Main Study
Number analyzed (Participants) | 109
log10 HIV-1 RNA copies per mL
  Change at Week 2: number analyzed (Participants) | 100
  Change at Week 2 | -1.65 (0.056)
  Change at Week 4: number analyzed (Participants) | 99
  Change at Week 4 | -2.02 (0.066)
  Change at Week 8: number analyzed (Participants) | 102
  Change at Week 8 | -2.43 (0.086)
  Change at Week 12: number analyzed (Participants) | 101
  Change at Week 12 | -2.78 (0.080)
  Change at Week 24: number analyzed (Participants) | 97
  Change at Week 24 | -3.08 (0.096)
  Change at Week 36: number analyzed (Participants) | 99
  Change at Week 36 | -3.14 (0.102)
  Change at Week 48: number analyzed (Participants) | 95
  Change at Week 48 | -3.14 (0.099)

3. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Week 24
Description: Percentage of participants with HIV-1 RNA < 50 copies/mL were reported.
Time Frame: Week 24
Population: The ITT analysis set included all the participants who were randomized and received at least one dose of study treatment in the study.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | D/C/F/TAF: Main Study
Number analyzed (Participants) | 109
Percentage of Participants | 81.7 [73.35 to 87.80]

4. Secondary Outcome: Change From Baseline in Cluster of Differentiation 4 (CD4+) Cell Count at Weeks 12, 24 and 48
Description: The immunologic change was determined by changes in Cluster of CD4+ cell count. Change from baseline in CD4+ cell count at Weeks 12, 24 and 48 were assessed.
Time Frame: Baseline, Weeks 12, 24 and 48
Population: The ITT analysis set included all the participants who were randomized and received at least one dose of study treatment in the study. Here, n (number analyzed) signifies participants analyzed for this OM at specified timepoints.
Measure: Mean (Standard Error); unit: Cells per millimeter cube (cells/mm^3)
Arm/Group | D/C/F/TAF: Main Study
Number analyzed (Participants) | 109
Cells per millimeter cube (cells/mm^3)
  Change at Week 12: number analyzed (Participants) | 100
  Change at Week 12 | 149.56 (16.621)
  Change at Week 24: number analyzed (Participants) | 96
  Change at Week 24 | 182.11 (16.885)
  Change at Week 48: number analyzed (Participants) | 94
  Change at Week 48 | 222.60 (20.618)

5. Secondary Outcome: Number of Participants That Required Discontinuation After Enrollment Based on Safety Stopping Rules
Description: Number of participants that required discontinuation after enrollment based on safety stopping rules were reported. Stopping rules include the following reasons: a). Estimated glomerular filtration rate (eGFR) according to the Modification of Diet in Renal Disease (MDRD) formula < 50 milliliter per minute (mL/min) b). Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) greater than or equal to (>=) 2.5*upper limit of normal (ULN); c). Serum lipase >=1.5*ULN; d). Positive serum human chorionic gonadotropin pregnancy test (beta-hCG) for women of childbearing potential; e). Laboratory results that the investigator believes should result in discontinuation of study medication; f). Participants identified with active hepatitis C virus (HCV) infection that in the opinion of the investigator requires HCV treatment immediately or expected to be needed during the course of the study with agents not compatible with D/C/F/TAF FDC.
Time Frame: Up to Week 48
Population: The safety analysis was performed on the ITT analysis set which included all enrolled participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | D/C/F/TAF: Main Study
Number analyzed (Participants) | 109
Participants | 3

6. Secondary Outcome: Percentage of Participants Discontinuing Therapy Due to Adverse Events (AEs)
Description: Percentage of participants discontinuing therapy due to AEs were reported. An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship.
Time Frame: Up to Week 48
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | D/C/F/TAF: Main Study
Number analyzed (Participants) | 109
Percentage of participants | 0.9

7. Secondary Outcome: Percentage of Participants Experiencing Grade 3 and 4 Adverse Events
Description: AE is any untoward medical occurrence in participant who received study drug without regard to possibility of causal relationship. Events with Grade 3 or higher (3=Severe; 4=life-threatening; 5=fatal) are events that significantly interrupt usual daily activity, require systemic drug therapy/other treatment and are, in many situations, considered unacceptable or intolerable events.
Time Frame: Up to Week 48
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | D/C/F/TAF: Main Study
Number analyzed (Participants) | 109
Percentage of participants
  Grade 3 | 11.9
  Grade 4 | 0.9

8. Secondary Outcome: Percentage of Participants Experiencing Grade 3 and 4 Laboratory Abnormalities
Description: Percentage of participants experiencing grade 3 and 4 laboratory abnormalities was assessed by Division of Acquired Immunodeficiency Syndrome (DAIDS) Adverse Event (AE) Grading Table. Abnormal laboratory values with Grade 3 or higher (3=Severe; 4=potentially life-threatening) signifies an interruption of usual daily activity, requiring systemic drug therapy/other treatment and are, in many situations, considered unacceptable or intolerable.
Time Frame: Up to Week 48
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | D/C/F/TAF: Main Study
Number analyzed (Participants) | 109
Percentage of participants
  ALT: Grade 3 | 0
  ALT: Grade 4 | 2.8
  AST: Grade 3 | 0.9
  AST: Grade 4 | 3.7
  Calcium: Grade 3 | 0
  Calcium: Grade 4 | 0.9
  Glucose: Grade 3 | 0.9
  Glucose: Grade 4 | 0
  Hyperbilirubinemia: Grade 3 | 2.8
  Hyperbilirubinemia: Grade 4 | 0
  Hypophosphatemia: Grade 3 | 0.9
  Hypophosphatemia: Grade 4 | 0
  Sodium: Grade 3 | 0
  Sodium: Grade 4 | 0.9
  Absolute Lymphocytes Count: Grade 3 | 0.9
  Absolute Lymphocytes Count: Grade 4 | 0.9
  Platelet Count: Grade 3 | 0
  Platelet Count: Grade 4 | 0.9

9. Secondary Outcome: Percentage of Participants Meeting Resistance Stopping Rules, Requiring Discontinuation of Study Treatment Due to Baseline Resistance Findings
Description: Percentage of participants meeting resistance stopping rules, requiring discontinuation of study treatment due to baseline resistance findings were reported. Investigator reviewed antiretroviral screening/baseline resistance data at Week 4, depending on availability of screening/baseline HIV genotypic drug resistance testing results from central laboratory. Participants who do not show full sensitivity to all drugs in the fixed-dose combination (FDC) study regimen according to the susceptibility assessment in the Genosure Prime report will be contacted to return to study site for early study treatment discontinuation (ESTD). Participants with identified resistance to lamivudine/Emtricitabine, attributed to the presence of the M184I/V mutation alone will be permitted to remain in the study.
Time Frame: Up to Day 35
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | D/C/F/TAF: Main Study
Number analyzed (Participants) | 109
Percentage of participants | 0

10. Secondary Outcome: Percentage of Participants With Baseline Protease (PI), Reverse Transcriptase (RT) and Integrase (INI)-Resistance-associated Mutation (RAMs)
Description: Percentage of Participants with resistance-associated mutations present at baseline were reported and included mutations in the domain of PR, RT (including nucleoside reverse transcriptase inhibitor [NRTIs] and non-nucleoside/nucleotide reverse transcriptase inhibitor [NNRTIs]), INI, RAMs as determined by the GenoSure Prime assay. Genotypes were not available for 7 participants due to failed amplification of viral deoxyribo nucleic acid (DNA) (that is, low viral load (VL) [<500 copies/mL], reduced viral fitness, compromised sample collection/handling, primer incompatibility).
Time Frame: Baseline (Day 1)
Population: The ITT analysis set included all the participants who were randomized and received at least one dose of study treatment in the study. Here, N (number of participants analyzed) signifies participants evaluated for this endpoint.
Measure: Number; unit: Percentage of Participants
Arm/Group | D/C/F/TAF: Main Study
Number analyzed (Participants) | 102
Percentage of Participants
  Primary PI RAM | 4.9
  Secondary PI RAM | 98.0
  Darunavir RAM | 0
  Emtricitabine RAM | 2.0
  NNRTI RAM | 27.5
  Primary INI RAM | 0
  Secondary INI RAM | 4.9

11. Secondary Outcome: Percentage of Participants With Protocol-defined Virologic Failure (PDVF) at Week 24 and 48
Description: Virologic failure is defined as: a) Virologic Nonresponse: HIV-1 RNA <1 log10 reduction from baseline, and HIV-1 RNA >= 400 copies/mL at the Week 12 visit, subsequently confirmed at an unscheduled visit conducted within 2 to 4 weeks after Week 12. b) Virologic Rebound: At any visit, after achieving confirmed consecutive HIV-1 RNA <50 copies/mL, a rebound in HIV 1 RNA to >= 50 copies/mL, which is subsequently confirmed at a scheduled or unscheduled visit conducted within 2 to 4 weeks of the HIV-1 RNA result; or At any visit, a >1 log10 increase in HIV-1 RNA from the nadir, which is subsequently confirmed at the following scheduled or unscheduled visit conducted within 2 to 4 weeks of the HIV-1 RNA result.
Time Frame: Week 24 and 48
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | D/C/F/TAF: Main Study
Number analyzed (Participants) | 109
Percentage of participants
  Week 24 | 0
  Week 48 | 0

12. Secondary Outcome: Percentage of Participants Developing Resistance-associated Mutation (RAMs) and Loss of Phenotypic Susceptibility, Upon Meeting Protocol-defined Virologic Failure (PDVF)
Description: Percentage of participants developing RAMs and loss of phenotypic susceptibility, upon meeting PDVF were reported. Virologic failure is defined as: a) Virologic Nonresponse: HIV-1 RNA <1 log10 reduction from baseline, and HIV-1 RNA greater than or equal to (>=) 400 copies/mL at the Week 12 visit, subsequently confirmed at an unscheduled visit conducted within 2 to 4 weeks after Week 12. b) Virologic Rebound: At any visit, after achieving confirmed consecutive HIV-1 RNA <50 copies/mL, a rebound in HIV 1 RNA to >= 50 copies/mL, which is subsequently confirmed at a scheduled or unscheduled visit conducted within 2 to 4 weeks of the HIV-1 RNA result; or At any visit, a >1 log10 increase in HIV-1 RNA from the nadir, which is subsequently confirmed at the following scheduled or unscheduled visit conducted within 2 to 4 weeks of the HIV-1 RNA result.
Time Frame: Up to Week 48
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | D/C/F/TAF: Main Study
Number analyzed (Participants) | 109
Percentage of participants | 0

13. Secondary Outcome: Percentage of Participants Lost-to-Follow-up Throughout the 48 Weeks of Treatment
Description: Percentage of participants lost-to-follow-up throughout the 48 Weeks of treatment were reported.
Time Frame: Up to Week 48
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | D/C/F/TAF: Main Study
Number analyzed (Participants) | 109
Percentage of participants | 3.67

14. Secondary Outcome: Percentage of Participants With Retention in Care Completed and With Documented Clinical Visit
Description: Percentage of participants with retention in care completed and with documented clinical visit (within 90 days of discontinuation) were reported.
Time Frame: Up to Week 48
Population: The modified ITT analysis set included all participants who were randomized and received at least one dose of study treatment and are HIV-1 positive after enrollment. Here, 'N' (number of participants analyzed) signifies participants who were evaluable for this OM. Here, n (number analyzed) signifies participants analyzed at specified categories.
Measure: Number; unit: Percentage of participants
Arm/Group | D/C/F/TAF: Main Study
Number analyzed (Participants) | 11
Percentage of participants
  Retention in care: Completed | 63.6
  Documented Clinical Visit: number analyzed (Participants) | 7
  Documented Clinical Visit | 85.7

15. Secondary Outcome: Percentage of Participants With Treatment Adherence >95% Based on Pill Count at Weeks 4, 8, 12, 24, 36, and 48
Description: Percentage of participants with treatment adherence >95% based on pill count at Weeks 4, 8, 12, 24, 36, and 48 were reported. Treatment adherence was defined as having a treatment adherence of greater than (>) 95 percent (%) by pill count.
Time Frame: Weeks 4, 8, 12, 24, 36, and 48
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | D/C/F/TAF: Main Study
Number analyzed (Participants) | 109
Percentage of participants
  >95% at Week 4 | 83.5
  >95% at Week 8: number analyzed (Participants) | 97
  >95% at Week 8 | 84.5
  >95% at Week 12: number analyzed (Participants) | 97
  >95% at Week 12 | 79.4
  >95% at Week 24: number analyzed (Participants) | 98
  >95% at Week 24 | 76.5
  >95% at Week 36: number analyzed (Participants) | 99
  >95% at Week 36 | 75.8
  >95% at Week 48: number analyzed (Participants) | 96
  >95% at Week 48 | 65.6

16. Secondary Outcome: Percentage of Participants With 100% Treatment Adherence Based on Participants Self-Report, Using a 4-Day Recall at Weeks 4, 8, 12, 24, 36, and 48
Description: Percentage of participants with 100 % adherence based on participants self-report, using a 4-Day recall at Weeks 4, 8, 12, 24, 36, and 48 was reported.
Time Frame: Weeks 4, 8, 12, 24, 36, and 48
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percentage of participants
Arm/Group | D/C/F/TAF: Main Study
Number analyzed (Participants) | 109
Percentage of participants
  Week 4: number analyzed (Participants) | 104
  Week 4 | 99.76 (2.440)
  Week 8: number analyzed (Participants) | 100
  Week 8 | 99.50 (3.518)
  Week 12: number analyzed (Participants) | 102
  Week 12 | 99.02 (6.967)
  Week 24: number analyzed (Participants) | 100
  Week 24 | 98.04 (10.949)
  Week 36: number analyzed (Participants) | 99
  Week 36 | 99.49 (3.535)
  Week 48: number analyzed (Participants) | 97
  Week 48 | 99.48 (3.571)

17. Secondary Outcome: Mean Total Scores for the HIV-Treatment Satisfaction Questionnaire (HIVTSQs) at Weeks 4, 24, and 48
Description: The HIV treatment satisfaction questionnaire (HIVTSQ) is based on a 10-item self-reported scale that measures overall satisfaction with treatment. The HIVTSQ items are summed up to produce a treatment satisfaction score (0 to 60) and an individual satisfaction rating for each item (0 to 6). The higher the score, the greater the treatment satisfaction.
Time Frame: Weeks 4, 24, and 48
Population: as for outcome 4
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | D/C/F/TAF: Main Study
Number analyzed (Participants) | 109
Units on a scale
  Week 4: number analyzed (Participants) | 103
  Week 4 | 56.52 (0.472)
  Week 24: number analyzed (Participants) | 100
  Week 24 | 57.87 (0.387)
  Week 48: number analyzed (Participants) | 96
  Week 48 | 57.88 (0.442)

18. Secondary Outcome: Number of Participants With Hospitalizations
Description: Number of participants with hospitalizations (overnight) was reported.
Time Frame: Up to Week 48
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | D/C/F/TAF: Main Study
Number analyzed (Participants) | 109
Participants | 11

19. Secondary Outcome: Duration of Hospitalizations
Description: Duration of hospitalizations in days was reported for those participants hospitalized during the course of the study. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this OM.
Time Frame: Up to Week 48
Population: as for outcome 3
Measure: Median (Full Range); unit: Days
Arm/Group | D/C/F/TAF: Main Study
Number analyzed (Participants) | 11
Days | 5.0 [1 to 15]

20. Secondary Outcome: Number of Participants With Outpatient Visits
Description: Number of participants with outpatient visits (in addition to study visits, including General practitioner visit, Specialist visit, Nurse practitioner visit, Physician assistant visit, Home healthcare nurse visit and Other visit) was reported.
Time Frame: Up to Week 48
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | D/C/F/TAF: Main Study
Number analyzed (Participants) | 109
Participants
  General practitioner visit | 33
  Specialist visit | 28
  Nurse practitioner visit | 16
  Physician assistant visit | 6
  Home healthcare nurse visit | 0
  Other visit | 25

21. Secondary Outcome: Number of Participants With Emergency Room Visits
Description: Number of participants with emergency room visits was reported.
Time Frame: Up to Week 48
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | D/C/F/TAF: Main Study
Number analyzed (Participants) | 109
Participants | 19

22. Secondary Outcome: Median Medical Costs of Care ((United States of America [USA] Dollars) Based on Healthcare Resource Utilization [HRU])
Description: Median medical costs of care (United States of America [USA] dollars) based on healthcare resource utilization [HRU]) were reported. The cost of care specified for overnight hospitalization, hospital day care ward (without overnight), emergency room visit, general practitioner visit, specialist visit, nurse practitioner visit, physician assistant visit and Other visit.
Time Frame: Up to Week 48
Population: The ITT analysis set included all the participants who were randomized and received at least one dose of study treatment in the study. Here, n (number analyzed) signifies those participants who were evaluable for the specified categories.
Measure: Median (Full Range); unit: USA dollars
Arm/Group | D/C/F/TAF: Main Study
Number analyzed (Participants) | 109
USA dollars
  Overnight hospitalization: number analyzed (Participants) | 11
  Overnight hospitalization | 2035.0 [2035 to 4070]
  Hospital day care ward (without overnight): number analyzed (Participants) | 1
  Hospital day care ward (without overnight) | 341.0 [341 to 341]
  Emergency room visit: number analyzed (Participants) | 19
  Emergency room visit | 212.0 [212 to 424]
  General practitioner visit: number analyzed (Participants) | 33
  General practitioner visit | 142.0 [71 to 355]
  Specialist visit: number analyzed (Participants) | 27
  Specialist visit | 94.0 [94 to 752]
  Nurse practitioner visit: number analyzed (Participants) | 16
  Nurse practitioner visit | 66.0 [66 to 264]
  Physician assistant visit: number analyzed (Participants) | 6
  Physician assistant visit | 47.0 [47 to 94]
  Other visit: number analyzed (Participants) | 25
  Other visit | 148.0 [16 to 788]

23. Secondary Outcome: Percentage of Participants Discontinuing Therapy Due to Adverse Events (AEs) Through Week 96
Description: as for outcome 6
Time Frame: Up to Week 96
Population: Safety analysis set (SAS) included all participants who received at least 1 dose of study drug and contributed any safety data after the start of study drug up to extension phase.
Measure: Number; unit: Percentage of participants
Groups:
- D/C/F/TAF: Extension Study: Participants who completed the Week 48 visit were given the opportunity to continue D/C/F/TAF treatment during the extension phase until the D/C/F/TAF FDC tablet became commercially available and was reimbursed, or could be accessed through another source, or until the sponsor terminated clinical development (Up to 96 Weeks).
Arm/Group | D/C/F/TAF: Extension Study
Number analyzed (Participants) | 80
Percentage of participants | 1.3

24. Secondary Outcome: Percentage of Participants Experiencing Grade 3 and 4 Adverse Events Through Week 96
Description: as for outcome 7
Time Frame: Up to Week 96
Population: as for outcome 23
Measure: Number; unit: Percentage of participants
Arm/Group | D/C/F/TAF: Extension Study
Number analyzed (Participants) | 80
Percentage of participants
  Grade 3 | 7.5
  Grade 4 | 2.5

25. Secondary Outcome: Percentage of Participants Experiencing Grade 3 and 4 Laboratory Abnormalities Through Week 96
Description: Percentage of participants experiencing grade 3 and 4 laboratory abnormalities were assessed by Division of Acquired Immunodeficiency Syndrome (DAIDS) Adverse Event (AE) Grading Table. Abnormal laboratory values with Grade 3 or higher (3=Severe; 4=potentially life-threatening) signifies an interruption of usual daily activity, requiring systemic drug therapy/other treatment and are, in many situations, considered unacceptable or intolerable.
Time Frame: Up to Week 96
Population: as for outcome 23
Measure: Number; unit: Percentage of participants
Arm/Group | D/C/F/TAF: Extension Study
Number analyzed (Participants) | 80
Percentage of participants
  Glucose: Grade 3 | 2.5
  Glucose: Grade 4 | 0
  Hypophosphatemia: Grade 3 | 1.3
  Hypophosphatemia: Grade 4 | 0

26. Secondary Outcome: Percentage of Participants With Protocol-defined Virologic Failure (PDVF) at Week 72 and 96
Description: as for outcome 11
Time Frame: Weeks 72 and 96
Population: Safety analysis set (SAS) included all participants who received at least 1 dose of study drug and contributed any safety data after the start of study drug up to extension phase. Here 'n' (number analyzed) signifies number of participants with observed virologic response at specified timepoints.
Measure: Number; unit: Percentage of participants
Arm/Group | D/C/F/TAF: Extension Study
Number analyzed (Participants) | 80
Percentage of participants
  Week 72: number analyzed (Participants) | 66
  Week 72 | 10.6
  Week 96: number analyzed (Participants) | 11
  Week 96 | 9.1

ADVERSE EVENTS:
Time Frame: Main study: Up to 48 Weeks; Extension Study: Up to 96 Weeks
Description: The safety analysis was performed on the Intent-to-treat analysis set (ITT) analysis set during main study (Week 0-48) included all the participants who were randomized and received at least one dose of study treatment in the study and safety analysis set (SAS) was used for the analyses during the extension study (Week 48-96) included all participants who received at least 1 dose of study drug and contributed any safety data after the start of study drug.
Arm/Group | D/C/F/TAF: Main Study | D/C/F/TAF: Extension Study
All-Cause Mortality (participants affected / at risk) | 0/109 | 0/80
Serious Adverse Events (participants affected / at risk) | 10/109 | 4/80
Other Adverse Events (participants affected / at risk) | 92/109 | 45/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | D/C/F/TAF: Main Study (N=109) | D/C/F/TAF: Extension Study (N=80)
Colitis (Gastrointestinal disorders) | 1 | 0
Pancreatitis Acute (Gastrointestinal disorders) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0
Abdominal Injury (Injury, poisoning and procedural complications) | 1 | 1
Muscle Rupture (Injury, poisoning and procedural complications) | 1 | 1
Road Traffic Accident (Injury, poisoning and procedural complications) | 1 | 0
Seizure (Nervous system disorders) | 1 | 0
Mania (Psychiatric disorders) | 1 | 0
Psychotic Disorder (Psychiatric disorders) | 1 | 0
Suicidal Ideation (Psychiatric disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Meningitis aseptic (Infections and infestations) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | D/C/F/TAF: Main Study (N=109) | D/C/F/TAF: Extension Study (N=80)
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Eosinophilia (Blood and lymphatic system disorders) | 2 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 6 | 3
Splenomegaly (Blood and lymphatic system disorders) | 1 | 1
Bradycardia (Cardiac disorders) | 1 | 1
Tachycardia (Cardiac disorders) | 2 | 0
Motion Sickness (Ear and labyrinth disorders) | 1 | 0
Goitre (Endocrine disorders) | 0 | 1
Hypogonadism (Endocrine disorders) | 1 | 1
Blindness Transient (Eye disorders) | 1 | 1
Lacrimation Increased (Eye disorders) | 1 | 0
Photophobia (Eye disorders) | 1 | 1
Photopsia (Eye disorders) | 1 | 1
Abdominal Discomfort (Gastrointestinal disorders) | 1 | 0
Abdominal Distension (Gastrointestinal disorders) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 3 | 3
Abdominal Pain Lower (Gastrointestinal disorders) | 2 | 0
Anogenital Dysplasia (Gastrointestinal disorders) | 1 | 1
Anorectal Discomfort (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 1
Dental Caries (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 27 | 5
Duodenogastric Reflux (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 3 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 0
Food Poisoning (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Lip Swelling (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 17 | 1
Paraesthesia Oral (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 3 | 0
Vomiting (Gastrointestinal disorders) | 10 | 1
Chest Discomfort (General disorders) | 1 | 0
Chest Pain (General disorders) | 1 | 0
Chills (General disorders) | 1 | 0
Fatigue (General disorders) | 7 | 2
Influenza Like Illness (General disorders) | 2 | 0
Malaise (General disorders) | 1 | 0
Non-Cardiac Chest Pain (General disorders) | 1 | 1
Oedema Peripheral (General disorders) | 1 | 0
Pain (General disorders) | 2 | 1
Peripheral Swelling (General disorders) | 0 | 1
Pyrexia (General disorders) | 6 | 0
Gallbladder Polyp (Hepatobiliary disorders) | 1 | 1
Hepatic Cyst (Hepatobiliary disorders) | 1 | 1
Hepatic Steatosis (Hepatobiliary disorders) | 1 | 1
Hepatotoxicity (Hepatobiliary disorders) | 1 | 1
Drug Hypersensitivity (Immune system disorders) | 1 | 1
Seasonal Allergy (Immune system disorders) | 2 | 0
Abscess (Infections and infestations) | 1 | 0
Abscess Limb (Infections and infestations) | 1 | 0
Acarodermatitis (Infections and infestations) | 1 | 0
Acute Hepatitis C (Infections and infestations) | 1 | 1
Acute Sinusitis (Infections and infestations) | 3 | 1
Anal Chlamydia Infection (Infections and infestations) | 4 | 3
Anorectal Human Papilloma Virus Infection (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 2 | 0
Cellulitis (Infections and infestations) | 1 | 0
Cellulitis Staphylococcal (Infections and infestations) | 1 | 0
Chlamydial Infection (Infections and infestations) | 4 | 1
Conjunctivitis (Infections and infestations) | 3 | 1
Conjunctivitis Viral (Infections and infestations) | 1 | 1
Cytomegalovirus Syndrome (Infections and infestations) | 1 | 0
Epididymitis (Infections and infestations) | 1 | 0
Folliculitis (Infections and infestations) | 1 | 1
Gastroenteritis Viral (Infections and infestations) | 3 | 0
Genitourinary Chlamydia Infection (Infections and infestations) | 1 | 0
Gonorrhoea (Infections and infestations) | 4 | 1
Hepatitis A (Infections and infestations) | 0 | 1
Herpes Zoster (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 3 | 0
Nasopharyngitis (Infections and infestations) | 4 | 1
Oral Herpes (Infections and infestations) | 1 | 0
Oropharyngeal Gonococcal Infection (Infections and infestations) | 1 | 1
Otitis Externa (Infections and infestations) | 1 | 0
Otitis Media (Infections and infestations) | 1 | 0
Papilloma Viral Infection (Infections and infestations) | 1 | 1
Periodontitis (Infections and infestations) | 1 | 1
Pharyngeal Chlamydia Infection (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 4 | 0
Pilonidal Cyst (Infections and infestations) | 1 | 0
Proctitis Gonococcal (Infections and infestations) | 4 | 1
Pyuria (Infections and infestations) | 1 | 0
Secondary Syphilis (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 2 | 1
Skin Infection (Infections and infestations) | 1 | 0
Syphilis (Infections and infestations) | 4 | 3
Tonsillitis (Infections and infestations) | 2 | 1
Tooth Infection (Infections and infestations) | 1 | 0
Tuberculosis (Infections and infestations) | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 5 | 3
Urinary Tract Infection (Infections and infestations) | 1 | 0
Viral Pharyngitis (Infections and infestations) | 1 | 0
Viral Upper Respiratory Tract Infection (Infections and infestations) | 1 | 0
Vulvovaginal Candidiasis (Infections and infestations) | 1 | 0
Anal Injury (Injury, poisoning and procedural complications) | 1 | 0
Exposure to Communicable Disease (Injury, poisoning and procedural complications) | 1 | 0
Human Bite (Injury, poisoning and procedural complications) | 1 | 0
Ligament Sprain (Injury, poisoning and procedural complications) | 2 | 0
Muscle Strain (Injury, poisoning and procedural complications) | 1 | 0
Post-Traumatic Neck Syndrome (Injury, poisoning and procedural complications) | 1 | 0
Procedural Pain (Injury, poisoning and procedural complications) | 2 | 0
Skin Laceration (Injury, poisoning and procedural complications) | 1 | 0
Blood Pressure Diastolic Increased (Investigations) | 1 | 0
Blood Pressure Increased (Investigations) | 3 | 1
Body Temperature Increased (Investigations) | 1 | 0
Cardiac Murmur (Investigations) | 1 | 0
Weight Decreased (Investigations) | 10 | 3
Weight Increased (Investigations) | 1 | 2
Abnormal Loss of Weight (Metabolism and nutrition disorders) | 3 | 1
Dyslipidaemia (Metabolism and nutrition disorders) | 1 | 1
Gout (Metabolism and nutrition disorders) | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 2 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0
Impaired Fasting Glucose (Metabolism and nutrition disorders) | 1 | 0
Increased Appetite (Metabolism and nutrition disorders) | 2 | 1
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 1 | 1
Vitamin D Deficiency (Metabolism and nutrition disorders) | 4 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 5 | 0
Cervical Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Flank Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Groin Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 | 4
Plantar Fasciitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Systemic Lupus Erythematosus (Musculoskeletal and connective tissue disorders) | 1 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 1
Tenosynovitis Stenosans (Musculoskeletal and connective tissue disorders) | 1 | 0
Trigger Finger (Musculoskeletal and connective tissue disorders) | 1 | 1
Adrenal Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Seborrhoeic Keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Vulvovaginal Warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Dizziness (Nervous system disorders) | 2 | 0
Headache (Nervous system disorders) | 10 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 1
Paraesthesia (Nervous system disorders) | 1 | 1
Seizure (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0
Abnormal Dreams (Psychiatric disorders) | 2 | 1
Adjustment Disorder (Psychiatric disorders) | 1 | 0
Adjustment Disorder with Depressed Mood (Psychiatric disorders) | 1 | 1
Adjustment Disorder with Mixed Anxiety and Depressed Mood (Psychiatric disorders) | 1 | 1
Alcoholic Hangover (Psychiatric disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 3 | 0
Bipolar Disorder (Psychiatric disorders) | 2 | 1
Depressed Mood (Psychiatric disorders) | 1 | 1
Depression (Psychiatric disorders) | 2 | 3
Drug Abuse (Psychiatric disorders) | 2 | 2
Initial Insomnia (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 5 | 2
Major Depression (Psychiatric disorders) | 1 | 1
Mental Status Changes (Psychiatric disorders) | 1 | 0
Panic Disorder (Psychiatric disorders) | 1 | 1
Psychotic Disorder (Psychiatric disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 1 | 1
Cervical Dysplasia (Reproductive system and breast disorders) | 3 | 2
Erectile Dysfunction (Reproductive system and breast disorders) | 3 | 3
Gynaecomastia (Reproductive system and breast disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 1
Dermal Cyst (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 4 | 1
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 1 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 1
Macule (Skin and subcutaneous tissue disorders) | 1 | 0
Night Sweats (Skin and subcutaneous tissue disorders) | 1 | 0
Pityriasis Rosea (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 4 | 1
Rash Macular (Skin and subcutaneous tissue disorders) | 2 | 0
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 2 | 0
Rash Papular (Skin and subcutaneous tissue disorders) | 1 | 0
Rash Pruritic (Skin and subcutaneous tissue disorders) | 1 | 0
Seborrhoea (Skin and subcutaneous tissue disorders) | 2 | 1
Skin Disorder (Skin and subcutaneous tissue disorders) | 1 | 0
Skin Hypopigmentation (Skin and subcutaneous tissue disorders) | 1 | 1
Diastolic Hypertension (Vascular disorders) | 1 | 0
Essential Hypertension (Vascular disorders) | 1 | 1
Flushing (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 8 | 3
Hypotension (Vascular disorders) | 1 | 0
Systolic Hypertension (Vascular disorders) | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1
Corneal abrasion (Injury, poisoning and procedural complications) | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Breast mass (Reproductive system and breast disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Study limitations included the open-label, single-arm study design and the small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2017-11-16): https://cdn.clinicaltrials.gov/large-docs/61/NCT03227861/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-18): https://cdn.clinicaltrials.gov/large-docs/61/NCT03227861/SAP_001.pdf